CLINICAL TRIAL: NCT02177773
Title: Evaluation of Gallium-68 DOTA-TOC Imaging of Somatostatin Receptor Positive Malignancies
Brief Title: GA-68 DOTA-TOC of Somatostatin Positive Malignancies
Acronym: DOTA-TOC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: FDA approved agent for this indication during enrollment
Sponsor: University of California, San Francisco (Other)
Collaborators: Peterson Family Foundation (Unknown)
Responsible Party: Principal Investigator, Thomas Hope, Assistant Professor of Radiology and Biomedical Engineering, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14453-HDFCCC; NCI-2017-00451 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Neuroendocrine Tumor; Paraganglioma; Carcinoid Tumors; Neuroblastoma
MeSH Terms: conditions — Neuroendocrine Tumors; Paraganglioma; Carcinoid Tumor; Neuroblastoma | interventions — gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga-68 DOTA-TOC PET/CT (Experimental): Patients receive Gallium Ga 68-DOTA-TOC IV over 1-2 minutes. Within 55-70 minutes, patients then undergo either a PET/CT scan lasting 30-40 minutes or a PET/MRI scan lasting 50 minutes.
  Interventions: Procedure: Computed Tomography (CT); Drug: Gallium Ga 68-Edotreotide; Procedure: Magnetic Resonance Imaging (MRI); Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Procedure: Computed Tomography (CT) — Undergo Gallium Ga 68-DOTA-TOC PET/CT
  Other Names: CAT; CAT Scan; Computed Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; Tomography
Drug: Gallium Ga 68-Edotreotide — Given Intravenously (IV) before imaging
  Other Names: Ga-68 DOTA0-Tyr3-octreotide; GALLIUM EDOTREOTIDE GA-68; Gallium Ga 68-DOTATOC
Procedure: Magnetic Resonance Imaging (MRI) — Undergo gallium Ga 68-DOTA-TOC PET/MRI
  Other Names: Magnetic Resonance Imaging; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography (PET) — Undergo gallium Ga 68-DOTA-TOC PET in combination with CT or MRI
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography; Positron Emission Tomography Scan; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
This phase I/II trial studies how well gallium Ga 68-DOTA-TOC positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI) works in imaging patients with somatostatin receptor positive tumors. Gallium Ga 68-DOTA-TOC binds to somatostatin receptor positive tumors and can be seen using a PET scan. A PET scan uses a special camera to detect energy given off from gallium Ga 68-DOTA-TOC, to make detailed pictures of areas where material accumulates in the body. Diagnostic procedures, such as gallium Ga 68-DOTA-TOC PET/CT or PET/MRI, may help find and diagnose somatostatin receptor positive tumors and help plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if gallium Ga 68-DOTA-TOC (gallium-68 labeled DOTA-TOC) results in the delineation of more lesions than with conventional imaging.

SECONDARY OBJECTIVES:

I. To determine if the incorporation of gallium (Ga)-68 DOTA-TOC PET/CT into the management decision making process results in a change in stage of the patient.

OUTLINE:

Patients receive gallium Ga 68-DOTA-TOC intravenously (IV) over 1-2 minutes. Within 55-70 minutes, patients then undergo a PET/CT scan over 30-40 minutes or a PET/MRI scan over 50 minutes.

After completion of study, patients are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected somatostatin receptor positive tumor such as carcinoid; neuroendocrine tumor; neuroblastoma; pheochromocytoma. Supporting evidence may include MRI, CT, biochemical markers, and or pathology report.
* Age > 1.
* Karnofsky performance status of > 50 (or Eastern Cooperative Oncology Group (ECOG) / World Health Organization (WHO) equivalent).
* Not pregnant. A negative serum pregnancy test is required for all female subjects with childbearing potential.
* Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

* Hepatic enzymes 5 times greater than the upper limits of normal, serum creatinine > 3.0 mg/dL (270 Micromole per liter (uM/L).
* Patients exceeding the weight limitations of the scanner or are not able to enter the bore of the PET /CT scanner due to BMI
* Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.); although at Mission Bay Hospital pediatric patients may be sedated per clinical protocol.
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.).
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study compliance.
* Recognized concurrent active infection Previous systemic or radiation treatment for another cancer of any type within the last 2 months.
* Use of any other investigational product or device within 30 days prior to dosing, or known requirement for any other investigational agent prior to completion of all scheduled study assessments

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DOTATOC Imaging: All patients received a single DOTATOC imaging study.
Period: Overall Study
Arm/Group | DOTATOC Imaging
Started | 300
Completed | 300
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ga-68 DOTA-TOC PET/CT: Patients receive gallium Ga 68-DOTA-TOC IV over 1-2 minutes. Within 55-70 minutes, patients then undergo a PET/CT scan over 30-40 minutes or a PET/MRI scan over 50 minutes.
  Computed Tomography: Undergo gallium Ga 68-DOTA-TOC PET/CT
  Gallium Ga 68-Edotreotide: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Magnetic Resonance Imaging: Undergo gallium Ga 68-DOTA-TOC PET/MRI
  Positron Emission Tomography: Undergo gallium Ga 68-DOTA-TOC PET/CT
  Positron Emission Tomography: Undergo gallium Ga 68-DOTA-TOC PET/MRI
Arm/Group | Ga-68 DOTA-TOC PET/CT
Number analyzed (Participants) | 300
Age, Customized [Count of Participants; unit: Participants]
  10-19 years | 2
  20-29 years | 6
  30-39 years | 22
  40-49 years | 38
  50-59 years | 71
  60-69 years | 106
  70-79 years | 48
  80-89 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 226
  Unknown or Not Reported | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 8
  White | 201
  More than one race | 2
  Unknown or Not Reported | 69
Region of Enrollment [Number; unit: participants]
  United States | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions as Determined by Gallium Ga 68-DOTA-TOC Positron Emission Tomography (PET) Imaging
Description: The 5 largest lesions in each of eight body regions (head and neck, mediastinum, lung, liver, pancreas, the remaining abdomen and pelvis, bone and lymph nodes), will be measured by size (short and long axis) as well as standardized uptake value maximum on conventional imaging and the gallium Ga 68-DOTA-TOC PET imaging. Additionally, the confidence that each lesion represents a metastasis will be recorded The five largest lesions will be (1 = benign, 2 = likely benign, 3 = indeterminant, 4 = likely malignant, 5 = malignant). The number of positive body regions using conventional imaging and Ga-68 DOTA-TOC PET/CT will be compared using a paired t-test (or Wilcoxon signed-rank test if the data appear to be non-normally distributed). The Wilcoxon signed-rank test will also be used to compare reader confidence of paired lesions between conventional imaging and Ga-68 DOTA-TOC PET/CT
Time Frame: 1 day
Population: Since the study agent was approved for the indication by FDA it was decided not to continue investigation and waste resources to analyze data collected to see if the agent is effective for the indication.
Arm/Group | DOTATOC Imaging
Number analyzed (Participants) | 0

2. Primary Outcome: Standardized Uptake Value Maximum (SUVmax)
Description: The 5 largest lesions in each of eight body regions (head and neck, mediastinum, lung, liver, pancreas, the remaining abdomen and pelvis, bone and lymph nodes), will be measured by size (short and long axis) as well as standardized uptake value maximum on conventional imaging and the gallium Ga 68-DOTA-TOC PET imaging. Additionally, the confidence that each lesion represents a metastasis will be recorded.
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | DOTATOC Imaging
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Clinical Stage as Determined by Conventional Imaging and Re-determined by Gallium Ga 68-DOTA-TOC PET Imaging
Description: Impact on care will be accessed for value added by the investigational Ga-68 DOTA-TOC PET/CT scan similar to assessment for impact on care as in the National Oncology PET registry. A percentage will then be calculated for both "Change in stage" with a 95% confidence interval determined.
Time Frame: Up to 2 weeks
Population: as for outcome 1
Arm/Group | DOTATOC Imaging
Number analyzed (Participants) | 0

4. Primary Outcome: Inter-reader Variability
Description: Inter-reader variability for the number of positive regions will be compared using Kappa statistics. In all cases we will provide point estimates and 95% confidence intervals for effects along with p-values.
Time Frame: 1 day
Population: as for outcome 1
Arm/Group | DOTATOC Imaging
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Two weeks
Description: All patients receiving Ga-68 DOTA-TOC were evaluated for safety. Safety parameters include physical findings and spontaneous reports of adverse events (AEs) reported to investigator by patients. Any grade 3 and above AEs were recorded. Patients were followed for two weeks after enrollment by phone, and all AEs were followed with appropriate medical management until resolved.
Arm/Group | DOTATOC Imaging
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 0/300

LIMITATIONS AND CAVEATS:
Since the study agent was approved for the indication by FDA it was decided not to continue investigation and waste resources to analyze data collected to see if the agent is effective for the indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-07-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT02177773/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT02177773/ICF_001.pdf